CLINICAL TRIAL: NCT01105533
Title: Phase I, Open-Label, Multi-Center, Accelerated Dose Escalation Study Of The Anti-Angiogenesis Agent PF-00337210 In Patients With Advanced Solid Tumors
Brief Title: A Dose Finding Study Of A New Medication, PF-00337210 That Will Possibly Decrease Blood Supply To Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8051001
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-02

CONDITIONS: Neoplasm
Keywords: VGEF inhibitor; Anti angiogenesis; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — PF 00337210

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Cohort 1 (Experimental)
  Interventions: Drug: PF-00337210
- Cohort 2 (Experimental)
  Interventions: Drug: PF-00337210
- Cohort 3 (Experimental)
  Interventions: Drug: PF-00337210
- Cohort 4 (Experimental)
  Interventions: Drug: PF-00337210
- Cohort 5 (Experimental)
  Interventions: Drug: PF-00337210
- Cohort 6 (Experimental)
  Interventions: Drug: PF-00337210
- Cohort 7 (Experimental)
  Interventions: Drug: PF-00337210
- Cohort 8 (Experimental)
  Interventions: Drug: PF-00337210
- Cohort 9 (Experimental)
  Interventions: Drug: PF-00337210
- Cohort 10 (Experimental)
  Interventions: Drug: PF-00337210

INTERVENTIONS:
Drug: PF-00337210 — 0.67mg Capsule Once Daily (Accelerated Dose Escalation) Continuous
  Arms: Cohort 1
Drug: PF-00337210 — 1mg Capsule Once Daily (Dose Escalation) Continuous
  Arms: Cohort 2
Drug: PF-00337210 — 2mg Capsule Once Daily (Dose Escalation) Continuous
  Arms: Cohort 3
Drug: PF-00337210 — 4mg Capsule Once Daily (Dose Escalation) Continuous
  Arms: Cohort 4
Drug: PF-00337210 — 6mg Capsule Once Daily (Dose Escalation) Continuous
  Arms: Cohort 5
Drug: PF-00337210 — 9mg Capsule Once Daily (Dose Escalation) Continuous
  Arms: Cohort 6
Drug: PF-00337210 — 8mg Capsule Once Daily (Dose Escalation) Continuous
  Arms: Cohort 7
Drug: PF-00337210 — 4mg Capsule Twice Daily (Dose Escalation) Continuous
  Arms: Cohort 8
Drug: PF-00337210 — 6mg Capsule Twice Daily (Dose Escalation) Continuous
  Arms: Cohort 9
Drug: PF-00337210 — 6mg Capsule Twice Daily (Dose Expansion) Continuous
  Arms: Cohort 10

SUMMARY:
This study will test a new cancer medication to determine if this medication will block blood supply to a tumor and decrease growth of a tumor. This study will also define the safety profile and define the safest dose of this new medication for people who have cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid tumors un-responsive to currently available therapies or for which there is no standard therapy.
* At least 1 measurable disease site as defined by Response Evaluation Criterion in Solid Tumors [RECIST].
* Adequate bone marrow, liver function and renal function as defined by protocol.
* Blood pressure Requirements During dose escalation - no evidence of pre-existing hypertension and no antihypertensive medications at baseline.

During dose expansion - patient's whose hypertension is controlled by antihypertensive therapy.

Exclusion Criteria:

* Chemotherapy, radiotherapy or any investigational therapy within 4 weeks of study entry
* Current use or anticipated need for drugs that are known CYP34 inhibitors or inducers.
* Patients with carcinomatous meningitis or un-treated brain metastases.
* Any acute cardiovascular incident within the past 12 months.
* Patients with active gastrointestinal bleeding or significant gastrointestinal abnormalities as defined by protocol
* Patients with no evidence of the following for 5 years: malignancy or metastatic disease of skin cancer (except melanoma), in situ cervical cancer or breast cancer or T1C prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-05; Primary Completion 2010-10 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8051001&StudyName=A%20Dose%20Finding%20Study%20Of%20A%20New%20Medication%2C%20PF-00337210%20That%20Will%20Possibly%20Decrease%20Blood%20Supply%20To%20Tumors%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-00337210 0.67 mg Once Daily: PF-00337210 0.67 milligram (mg) capsule orally once daily in cycles of 28 days.
- PF-00337210 1 mg Once Daily: PF-00337210 1 mg capsule orally once daily in cycles of 28 days.
- PF-00337210 2 mg Once Daily: PF-00337210 2 mg capsule orally once daily in cycles of 28 days.
- PF-00337210 4 mg Once Daily: PF-00337210 4 mg capsule orally once daily in cycles of 28 days.
- PF-00337210 6 mg Once Daily: PF-00337210 6 mg capsule orally once daily in cycles of 28 days.
- PF-00337210 8 mg Once Daily: PF-00337210 8 mg capsule orally once daily in cycles of 28 days.
- PF-00337210 9 mg Once Daily: PF-00337210 9 mg capsule orally once daily in cycles of 28 days.
- PF-00337210 4 mg Twice Daily: PF-00337210 4 mg capsule orally twice daily in cycles of 28 days.
- PF-00337210 6 mg Twice Daily: PF-00337210 6 mg capsule orally twice daily in cycles of 28 days.
Period: Overall Study
Arm/Group | PF-00337210 0.67 mg Once Daily | PF-00337210 1 mg Once Daily | PF-00337210 2 mg Once Daily | PF-00337210 4 mg Once Daily | PF-00337210 6 mg Once Daily | PF-00337210 8 mg Once Daily | PF-00337210 9 mg Once Daily | PF-00337210 4 mg Twice Daily | PF-00337210 6 mg Twice Daily
Started | 1 | 1 | 3 | 3 | 7 | 7 | 8 | 4 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 3 | 7 | 7 | 8 | 4 | 12
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 3 | 3 | 4 | 5 | 3 | 2 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-00337210: PF-00337210 0.67 mg, 1 mg, 2 mg, 4 mg, 6 mg, 8 mg or 9 mg capsule orally once daily or PF-00337210 4 mg or 6 mg capsule twice daily in cycles of 28 days.
Arm/Group | PF-00337210
Number analyzed (Participants) | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 53.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs included events occurring in Cycle 1: blood pressure of 180/110 millimeters of mercury (mmHg) or higher for 3 readings over 3 hours regardless of use of anti-hypertensive drugs or greater than (>) 160/100 mmHg for 3 readings over 3 days on maximum anti-hypertensive drugs; afebrile Grade 4 neutropenia for greater than or equal to (>=) 7 days or >=Grade 3 neutropenia associated with fever (1 reading of oral temperature >38.5 degree Celsius [degree C] or 3 readings of oral temperature >38.0 degree C in 24-hour period); Grade 4 thrombocytopenia; hemoptysis of >1/2 teaspoon of bright red blood per day; proteinuria of >=2 grams/24 hours; inability to resume PF-00337210 dosing at current dose level within 14 days of stopping due to treatment-related toxicity; >=Grade 3 nonhematological toxicities (except alopecia and blood pressure/hypertension); Grade 3 nonhematological toxicities that could be controlled to Grade 2 or less with appropriate treatment were not considered dose limiting.
Time Frame: Baseline up to Day 28
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | PF-00337210 0.67 mg Once Daily | PF-00337210 1 mg Once Daily | PF-00337210 2 mg Once Daily | PF-00337210 4 mg Once Daily | PF-00337210 6 mg Once Daily | PF-00337210 8 mg Once Daily | PF-00337210 9 mg Once Daily | PF-00337210 4 mg Twice Daily | PF-00337210 6 mg Twice Daily
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 6 | 5 | 4 | 12
participants | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD: dose level at which no more than 1 of 6 participants experienced DLT during Cycle 1. DLTs: blood pressure of 180/110 mmHg or higher for 3 readings over 3 hours regardless of use of anti-hypertensive drugs or >160/100 mmHg for 3 readings over 3 days on maximum anti-hypertensive drugs; afebrile Grade 4 neutropenia >=7 days or >= Grade 3 neutropenia associated with fever (1 reading of oral temperature >38.5 degree C or 3 readings of oral temperature >38.0 degree C in 24-hour period); Grade 4 thrombocytopenia; hemoptysis of >1/2 teaspoon of bright red blood per day; proteinuria of >=2 grams/24 hours; inability to resume PF-00337210 dosing at current dose level within 14 days of stopping due to treatment-related toxicity; >=Grade 3 nonhematological toxicities (except alopecia and blood pressure/hypertension); Grade 3 nonhematological toxicities that could be controlled to Grade 2 or less with appropriate treatment were not considered dose limiting.
Time Frame: Day 28
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: mg once daily
Arm/Group | PF-00337210
Number analyzed (Participants) | 46
mg once daily | 8

3. Primary Outcome: Maximum Administered Dose (MAD)
Description: MAD: dose level at which 2 or more out of 6 participants experienced DLT during Cycle 1. DLTs: blood pressure of 180/110 mmHg or higher for 3 readings over 3 hours regardless of use of anti-hypertensive drugs or >160/100 mmHg for 3 readings over 3 days on maximum anti-hypertensive drugs; afebrile Grade 4 neutropenia >=7 days or >= Grade 3 neutropenia associated with fever (1 reading of oral temperature >38.5 degree C or 3 readings of oral temperature >38.0 degree C in 24-hour period); Grade 4 thrombocytopenia; hemoptysis of >1/2 teaspoon of bright red blood per day; proteinuria of >=2 grams/24 hours; inability to resume PF-00337210 dosing at current dose level within 14 days of stopping due to treatment-related toxicity; >=Grade 3 nonhematological toxicities (except alopecia and blood pressure/hypertension); Grade 3 nonhematological toxicities that could be controlled to Grade 2 or less with appropriate treatment were not considered dose limiting.
Time Frame: Day 28
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: mg once daily
Arm/Group | PF-00337210
Number analyzed (Participants) | 46
mg once daily | 9

4. Primary Outcome: Recommended Phase-2 Dose (RP2D)
Description: RP2D was determined based on the safety profile and pharmacodynamic findings. The twice daily dosing was preferred over once daily dosing for RP2D, as per investigator's discretion, due to more consistent changes in pharmacodynamic markers and greater clinical benefit observed in twice daily dosing.
Time Frame: Day 28
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: mg twice daily
Arm/Group | PF-00337210
Number analyzed (Participants) | 46
mg twice daily | 6

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Pre-dose,0.5,1,2,4,6,8,10,16,20,24 hours(hrs) post-dose on Day 1(0.67 mg group);pre-dose,0.5,1,2,4,6,8,18,20,24 hrs post-dose on Day 1,15,29(once daily groups);pre-dose,0.5,1,2,4,6,8 hrs post-dose on Day 1,15,29 (twice daily groups);pre-dose on Day 43, 57
Population: Formal quality-assured, quality-controlled, pharmacokinetic (PK) analysis was not performed and hence, Cmax was not calculated.
Arm/Group | PF-00337210 0.67 mg Once Daily | PF-00337210 1 mg Once Daily | PF-00337210 2 mg Once Daily | PF-00337210 4 mg Once Daily | PF-00337210 6 mg Once Daily | PF-00337210 8 mg Once Daily | PF-00337210 9 mg Once Daily | PF-00337210 4 mg Twice Daily | PF-00337210 6 mg Twice Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose,0.5,1,2,4,6,8,10,16,20,24 hrs post-dose on Day 1(0.67 mg group);pre-dose,0.5,1,2,4,6,8,18,20,24 hrs post-dose on Day 1,15,29(once daily groups);pre-dose,0.5,1,2,4,6,8 hrs post-dose on Day 1,15,29 (twice daily groups);pre-dose on Day 43, 57
Population: Formal quality-assured, quality-controlled, pharmacokinetic (PK) analysis was not performed and hence, t1/2 was not calculated.
Arm/Group | PF-00337210 0.67 mg Once Daily | PF-00337210 1 mg Once Daily | PF-00337210 2 mg Once Daily | PF-00337210 4 mg Once Daily | PF-00337210 6 mg Once Daily | PF-00337210 8 mg Once Daily | PF-00337210 9 mg Once Daily | PF-00337210 4 mg Twice Daily | PF-00337210 6 mg Twice Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)]
Description: AUC (0-24)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-24).
Time Frame: as for outcome 6
Population: Formal quality-assured, quality-controlled, pharmacokinetic (PK) analysis was not performed and hence, AUC (0-24) was not calculated.
Arm/Group | PF-00337210 0.67 mg Once Daily | PF-00337210 1 mg Once Daily | PF-00337210 2 mg Once Daily | PF-00337210 4 mg Once Daily | PF-00337210 6 mg Once Daily | PF-00337210 8 mg Once Daily | PF-00337210 9 mg Once Daily | PF-00337210 4 mg Twice Daily | PF-00337210 6 mg Twice Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 6
Population: Formal quality-assured, quality-controlled, pharmacokinetic (PK) analysis was not performed and hence, AUC (0 - ∞) was not calculated.
Arm/Group | PF-00337210 0.67 mg Once Daily | PF-00337210 1 mg Once Daily | PF-00337210 2 mg Once Daily | PF-00337210 4 mg Once Daily | PF-00337210 6 mg Once Daily | PF-00337210 8 mg Once Daily | PF-00337210 9 mg Once Daily | PF-00337210 4 mg Twice Daily | PF-00337210 6 mg Twice Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Apparent Volume of Distribution (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose is influenced by the fraction absorbed.
Time Frame: as for outcome 6
Population: Formal quality-assured, quality-controlled, pharmacokinetic (PK) analysis was not performed and hence, Vss was not calculated.
Arm/Group | PF-00337210 0.67 mg Once Daily | PF-00337210 1 mg Once Daily | PF-00337210 2 mg Once Daily | PF-00337210 4 mg Once Daily | PF-00337210 6 mg Once Daily | PF-00337210 8 mg Once Daily | PF-00337210 9 mg Once Daily | PF-00337210 4 mg Twice Daily | PF-00337210 6 mg Twice Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Systemic Clearance (CL)
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 6
Population: Formal quality-assured, quality-controlled, PK analysis was not performed and hence, CL was not calculated.
Arm/Group | PF-00337210 0.67 mg Once Daily | PF-00337210 1 mg Once Daily | PF-00337210 2 mg Once Daily | PF-00337210 4 mg Once Daily | PF-00337210 6 mg Once Daily | PF-00337210 8 mg Once Daily | PF-00337210 9 mg Once Daily | PF-00337210 4 mg Twice Daily | PF-00337210 6 mg Twice Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Objective Response of Complete Response or Partial Response
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR defined as disappearance of all target and non-target lesions and no appearance of new lesions. Confirmed PR defined as at least 30 percent decrease in sum of the longest dimensions (LD) of the target lesions, taking as a reference the baseline sum LD, without progression of non-target lesions and no appearance of new lesions. Confirmed responses are those that persist on repeat imaging study >=4 weeks after initial documentation of response.
Time Frame: Baseline, every 8 weeks up to Cycle 25 (Week 100)
Population: Full Analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-00337210
Number analyzed (Participants) | 46
participants | 2

12. Secondary Outcome: Change From Baseline in Biomarkers at Day 1 of Each Cycle up to Cycle 25
Description: Biomarkers included soluble plasma proteins associated with angiogenesis (vascular endothelial growth factor [VEGF], soluble vascular endothelial growth factor-2 receptor [sVEGFR2], soluble vascular endothelial growth factor-3 receptor [sVEGFR3], soluble beta type platelet-derived growth factor [sPDGFR beta]) and tumor proliferation (soluble stem-cell factor receptor [sKIT])
Time Frame: Baseline, Day 1 of Cycle 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25
Population: Results are not reported as the data were not statistically summarized but available in individual participant listing.
Arm/Group | PF-00337210 0.67 mg Once Daily | PF-00337210 1 mg Once Daily | PF-00337210 2 mg Once Daily | PF-00337210 4 mg Once Daily | PF-00337210 6 mg Once Daily | PF-00337210 8 mg Once Daily | PF-00337210 9 mg Once Daily | PF-00337210 4 mg Twice Daily | PF-00337210 6 mg Twice Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Other Pre Specified Outcome: Effect of Food on Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)]
Description: as for outcome 7
Time Frame: Pre-dose,0.5,1,2,4,6,8,18,20,24 hrs post-dose on Day 29 (fasted state), Day 30 (fed state) for once daily groups, pre-dose,0.5,1,2,4,6,8 hrs post-dose on Day 29 Day 29 (fasted state), Day 30 (fed state) for twice daily groups
Population: Formal quality-assured, quality-controlled, PK analysis was not performed and hence, food effect on AUC (0-24) was not assessed.
Arm/Group | PF-00337210 0.67 mg Once Daily | PF-00337210 1 mg Once Daily | PF-00337210 2 mg Once Daily | PF-00337210 4 mg Once Daily | PF-00337210 6 mg Once Daily | PF-00337210 8 mg Once Daily | PF-00337210 9 mg Once Daily | PF-00337210 4 mg Twice Daily | PF-00337210 6 mg Twice Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-00337210
Serious Adverse Events (participants affected / at risk) | 19/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00337210 (N=46)
Leukocytosis (Blood and lymphatic system disorders) | 1
Polycythaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Disease progression (General disorders) | 4
Fatigue (General disorders) | 2
Pain (General disorders) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Electrocardiogram abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00337210 (N=46)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Palpitations (Cardiac disorders) | 2
Ear congestion (Ear and labyrinth disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Ear disorder (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Periorbital oedema (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 10
Abdominal pain lower (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 2
Anal haemorrhage (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 18
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 8
Eructation (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 18
Oesophageal pain (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Tongue exfoliation (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Chest discomfort (General disorders) | 3
Chest pain (General disorders) | 6
Chills (General disorders) | 5
Early satiety (General disorders) | 1
Fatigue (General disorders) | 23
Feeling cold (General disorders) | 1
Induration (General disorders) | 1
Localised oedema (General disorders) | 1
Mucosal inflammation (General disorders) | 2
Oedema (General disorders) | 3
Pain (General disorders) | 3
Pyrexia (General disorders) | 6
Bile duct obstruction (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Multiple allergies (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Eye injury (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wound necrosis (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 8
Band neutrophil count increased (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Blood alkaline phosphatase (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 2
Blood calcium decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Blood magnesium decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
Carbon dioxide decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Eosinophil count increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 3
International normalised ratio increased (Investigations) | 1
Monocyte count increased (Investigations) | 1
Neutrophil count (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Neutrophil count increased (Investigations) | 1
Troponin I increased (Investigations) | 1
Weight decreased (Investigations) | 8
White blood cell count (Investigations) | 1
White blood cell count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypophagia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 10
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Joint warmth (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 9
Dyskinesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 9
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Post herpetic neuralgia (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 2
Sensory disturbance (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 11
Urine odour abnormal (Renal and urinary disorders) | 1
Urogenital haemorrhage (Renal and urinary disorders) | 1
Breast discomfort (Reproductive system and breast disorders) | 1
Breast disorder (Reproductive system and breast disorders) | 1
Ejaculation disorder (Reproductive system and breast disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Blood blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 7
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Skin nodule (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 3
Hot flush (Vascular disorders) | 6
Hypertension (Vascular disorders) | 24
Phlebitis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Designation of outcomes as primary and secondary was based on study team input as study did not specify primary or secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.